CLINICAL TRIAL: NCT04783493
Title: Transcutaneous Magnetic Spinal Cord Stimulation for Freezing of Gait in Parkinson's Disease
Acronym: TMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USaoPaulo
Record Dates: First submitted 2021-02-22; First posted 2021-03-05 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Study is a randomized, double-blind, placebo-controlled, parallel, phase II clinical trial
Who Masked: Participant, Investigator
Masking Description: The random sequence will be generated by a computer program (randomization.com) using randomly exchanged blocks (size of four per block, active ratio / placebo 1: 1). Randomization will be stratified according to the severity of symptoms (TUG> 33 seconds = severe group; TUG ≤ 33 seconds = light group). The researchers will be specifically instructed not to break the randomization schedule in any way. Different researchers will carry out randomization, clinical evaluation and stimulation. Patients will be blinded to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE (Active Comparator): In the active group, non-invasive transcutaneous magnetic stimulation of the dorsal spine will be applied by placing a circular magnetic coil (Magventure®️ MagPro®️ R20) on the skin, in the upper thoracic region (chest level T2-T3). The stimulation intensity will represent 100% of the motor threshold, this determined by abdominal muscle contractions, found from single pulses, applied gradually every 10 seconds until the contractions appear. The intermittent theta burst stimulation protocol will consist of 20 stimulation trains, with an interval of 8 seconds between trains, each train will have 20 bursts, and each burst will have 3 pulses at 50 Hz repeated at 5 Hz. In total, 1200 pulses will be applied for 3 minutes and 58 seconds.
  Interventions: Device: Non-invasive magnetic stimulation of the spinal cord
- PLACEBO (Placebo Comparator): In the placebo group, a coil will be allocated in the T2-T3 thoracic region, however this coil will not be connected to the stimulation device, and another active coil will be positioned about 15cm behind, far from its field of view, to provide idea from the sound stimulus that is being stimulated. To create a sensation of muscle contraction and impression of active stimulation, both the placebo and active groups will be subjected to the sensory effect of transcutaneous electrical neurostimulation (TENS).
  Interventions: Other: Coil will not be connected to the stimulation device

INTERVENTIONS:
Device: Non-invasive magnetic stimulation of the spinal cord — Non-invasive transcutaneous magnetic stimulation of the dorsal spine will be applied by placing a circular magnetic coil (Magventure®️ MagPro®️ R20) on the skin, in the upper thoracic region (chest level T2-T3). The stimulation intensity will represent 100% of the motor threshold. The intermittent theta burst stimulation protocol will consist of 20 stimulation trains, with an interval of 8 seconds between trains, each train will have 20 bursts, and each burst will have 3 pulses at 50 Hz repeated at 5 Hz. In total, 1200 pulses will be applied for 3 minutes and 58 seconds
  Other Names: TMS
  Arms: ACTIVE
Other: Coil will not be connected to the stimulation device — coil will not be connected to the stimulation device, and another active coil will be positioned about 15cm behind, far from its field of view, to provide idea from the sound stimulus that is being stimulated
  Arms: PLACEBO

SUMMARY:
Dopaminergic drugs partially alleviate gait problems in Parkinson's disease, but the effects are not sustained in the long-term. Particularly, the freezing of gait, balance problems and other gait issues directly impacts patients' quality of life. Experimental epidural spinal cord stimulation studies have suggested positive effects on locomotion among PD patients, but the effects of non invasive stimulation have never been explored.

DETAILED DESCRIPTION:
The present study is a randomized, double-blind, placebo-controlled, parallel, phase II clinical trial that will assess the efficacy and safety of transcutaneous magnetic spinal cord stimulation in PD patients who have gait and balance changes refractory to dopaminergic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (not pregnant) aged between 21 and 80 years old;
2. Participants with idiopathic Parkinson's disease in Hoehn Yahr stages between 2 and 4 (moderate disease) during off-medication, whose primary symptom includes change in gait and / or balance (score equal to or greater than 1 in subitem 2.12 of the MSD scale -UPDRS ["gait and balance"]). The participant must also present freezing (block) of gait (score equal to or greater than 1 in sub-item 2.13 of the MSD-UPDRS scale - "freezing"). Patients should experience the above symptoms even though they are optimized from the medication point of view. The criteria for being optimized will be defined by a neurologist specialized in movement disorders who will evaluate the case. The presence of freezing will be confirmed through a specific scale (FOG score).
3. Mini-examination of mental status greater than or equal to 24 points;
4. Able to give informed consent in accordance with institutional policies;
5. Able to meet all testing and monitoring requirements, as defined by the study protocol;

Exclusion Criteria:

1. Patients with unstabilized psychiatric comorbidities
2. Impossibility to consent to your participation in the study.
3. Patients with uncontrolled infection or other pre-existing uncontrolled medical conditions (eg, decompensated diabetes, high blood pressure, pneumo or symptomatic heart disease).
4. Concomitant treatment with other experimental drugs.
5. Pregnant or breastfeeding women.
6. Presence of chronic pain in the lower limbs.
7. Patients who are unable to walk without assistance (cane, crutch, walker) or help from another person when they are without their medications for Parkinson's disease (off-medication).

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-29 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
TUG | Post-stimulation: immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  The primary outcome will be the change in gait speed between pre-stimulation and post-stimulation conditions between the two groups (active and placebo) assessed using the 5-meter total Timed Up and Go Test (TUG). Mixel model ANOVA, with TUG as the dependent variable, and time and group as independent variables -'group' would have two levels ('active' and 'placebo'). Our alternative hypothesis is that 'the time vs. group' interaction effect is significant. Then we should use post hoc statistical tests to explore our data further and to compare the effects of active versus placebo at different time levels.

SECONDARY OUTCOMES:
Secondary outcomes will be the change on other gait measures, gait speed. | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Evaluate the gait speed through measurements obtained through sensors for gait, during the gait of five meters.
Secondary outcomes will be the effects of stimulation on other gait measures, step length, stride length and step width. | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Evaluate step length, stride length and step width through measurements obtained through sensors for gait, during the gait of five meters.
Secondary outcomes will be the effects of stimulation on other gait measures, cadencia. | Baseline, immediately after the fifth day of stimulation, seven days after finishing the stimulation, twenty-eight days after finishing the stimulation.
  Evaluate the cadencia through measurements obtained through sensors for gait, during the gait of five meters.
Secondary outcomes will be the effects of stimulation on balance after noninvasive magnetic stimulation of the dorsal spine in patients with parkinson's disease. | Baseline, seven days after finishing the stimulation, twenty-eight days after finishing the stimulation.
  Evaluate the improvement of the balance through the application of questionnaires,which will be the Activities-specific Balance Confidence Scale (ABC) and Falls Efficacy Scale (FES I).
Determination of possible adverse effects of noninvasive magnetic stimulation of the dorsal spine in patients with parkinson's disease. | Immediately after the fifth day of stimulation, seven days after finishing the stimulation, twenty-eight days after finishing the stimulation.
  The patient will be actively questioned about the appearance of adverse effects of noninvasive stimulation of the dorsal cord.
Assess the effects of transcutaneous magnetic stimulation of the dorsal cord on quality of life in patients with parkinson's disease | Baseline, seven days after finishing the stimulation, twenty-eight days after finishing the stimulation.
  The questionnaire Parkinson Disease Questionnaire-39 (PDQ-39) will be applied.
To evaluate the effects of noninvasive stimulation of the dorsal cord in the presence of freezing gait, through the application of questionnaires. | Baseline, immediately after the fifth day of stimulation, seven, fourteen, twenty-one and twenty-eight days after finishing the stimulation.
  The questionnaires New Freezing of Gait Questionnaire (NFOG-Q), Sub-items 2.12 and 2.13 MDS-UPDRS will be applied.
Assess the effects of transcutaneous magnetic stimulation of the spinal cord on the other motor symptoms of Parkinson's disease. | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Other motor effects will be assessed by applying the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) item III and FOG SCORE.
Assess the effects of transcutaneous magnetic stimulation of the spinal cord on cognition of Parkinson's disease. | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Possible changes in cognition will be assessed based on the application of the Frontal assessment battery (FAB).

CONTACTS AND LOCATIONS:
Overall Officials: Rubens G Cury, MD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
WE CURRENTLY PLACE STUDY DATA ON THE REDCAP PLATFORM